CLINICAL TRIAL: NCT03527576
Title: Block Duration After Spinal Block and iv Dexamethasone: a Randomized Controlled Double-blinded Trial
Brief Title: Block Duration After Spinal Block and iv Dexamethasone.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2018-00500
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain; Lower Limb Injury
MeSH Terms: conditions — Pain, Postoperative; Leg Injuries | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): Intravenous injection of 0.15 mg/kg of dexamethasone before the surgery.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Intravenous injection of NaCl 0,9% before the surgery.
  Interventions: Drug: NaCl 0.0308 MEQ/ML Injectable Solution

INTERVENTIONS:
Drug: Dexamethasone — Intravenous injection of 0.15 mg/kg of dexamethasone before the surgery.
  Arms: Dexamethasone
Drug: NaCl 0.0308 MEQ/ML Injectable Solution — Intravenous injection of NaCl 0.9% before the surgery.
  Arms: Placebo

SUMMARY:
It has been largely demonstrated that iv dexamethasone prolongs the duration of analgesia after peripheral nerve block. However, data are missing regarding the duration of analgesia after spinal block. The objective of this randomized controlled double-blinded trial is to assess whether intravenous dexamethasone administered after a spinal block, before the surgery would prolong sensory block characteristics without impacting the motor block duration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ASA I-III status ;
* Patient scheduled for an osteosynthesis surgy of the lower limb

Exclusion Criteria:

* Polytrauma patient
* Pregnancy
* Contraindication to spinal anesthesia
* Contraindication to dexamethasone administration
* Patient with chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block (minutes) | Postoperative day 0
  Time interval between injection of the local anaesthetic and the regression of 2 dermatoma, compared to the highest dermatoma reached

SECONDARY OUTCOMES:
Highest dermatoma reached (level) | Postoperative day 0
Onset time between injection and highest dermatoma (minutes) | Postoperative day 0
Total duration of the sensory block (minutes) | Postoperative day 0
Total duration of the motor block (minutes) | Postoperative day 0
Time to the first analgesic request (minutes) | Postoperative day 0
Cumulative consumption of morphine (mg) | Postoperative days 0, 1 and 2
Pain score | Postoperative days 0, 1 and 2
  Numeric rating scale (0-10)
Rate of postoperative nausea and vomiting | Postoperative day 0, 1 and 2
  YES/NO
Rate of pruritus | Postoperative day 0, 1 and 2
  YES/NO
Rate of urinary retention | Postoperative day 1 and 2
  YES/NO
Satisfaction level | Postoperative day 2
  Numeric rating scale (0-10)
Length of stay | up to 14 days
  Days
Persistent pain | 3 and 6 postoperative months
  YES/NO
Pain score if persistent pain | 3 and 6 postoperative months
  Numeric rating scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bikfalvi A, Hofmann G, Bashawyah A, Rossel JB, Gonvers E, Albrecht E. Sensory block duration after spinal anaesthesia supplemented with intravenous dexamethasone: a randomised controlled double-blinded trial. Br J Anaesth. 2023 Jun;130(6):780-785. doi: 10.1016/j.bja.2023.02.027. Epub 2023 Mar 23. PMID 36966023